14 August 2018

Sponsor: Harvard University

Investigator: Adam Jaroszewski, A.M.

Randomized Controlled Trial of an Online Machine Learning-Driven Risk Assessment and Intervention Platform for Increasing the Use of Crisis Services

Statistical Analysis Plan

## Statistical Analysis Plan

We used chi-square tests to determine whether the treatment and control groups were equivalent on baseline factors (e.g., suicidal thoughts/behaviors). We conducted a chi-square test to examine the hypothesis that individuals assigned to the intervention condition would report using crisis resources at higher rates than individuals in the control condition. We used a chi-square test to determine whether individuals assigned to the intervention condition would rate their experience using Koko as "good" at higher rates than individuals in the control condition. Follow-up analyses consisted of a chi-square test to examine whether groups differed in terms of which crisis resource they used and a series of logistic regressions to examine potential moderators (e.g., history of suicidal thoughts/behavior, risk level) of the effect of intervention on the rate of using crisis resources.